CLINICAL TRIAL: NCT01704664
Title: Prospective Study of the Effect of Perioperative Immunonutrition on the Immune Host Defense and the Phagocytic and Bactericidal Activity of Blood Platelets in Gastric Cancer Patients.
Brief Title: Perioperative Immunonutrition, Phagocytic and Bactericidal Activity of Blood Platelets in Gastric Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3-37878 L
Record Dates: First submitted 2012-09-26; First posted 2012-10-11 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Gastric Cancer
Keywords: malnutrition,; perioperative artificial nutrition,; immunonutrition,; gastrectomy,; lymphocytes,; interleukin,; blood platelets,; phagocytic and bactericidal activity of blood platelets
MeSH Terms: conditions — Stomach Neoplasms; Malnutrition | interventions — Glutamine; Arginine; alanylglutamine; fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I - Nutritional therapy only during the postoperative period. (Active Comparator): Postoperative nutritional therapy administered in group I will not include immunomodulating factors. Early postoperative enteral nutrition, based on standard elementary diet (Peptisorb), starts 20 hours post-surgery. The initial flow rate will be 8 ml/h, which will be increased gradually, with the volume doubled every 24 hours, up to 100 ml/h. The enteral nutrition will be continued for six days. During the initial five days post-surgery, the patients will be additionally supplemented parenterally via peripheral veins (commercially available two-chamber bag for peripheral access with 480 kcal of energetic value and 5.7g of N contained in standard amino acids).
  Interventions: Dietary Supplement: Early postoperative enteral nutrition, based on standard elementary diet (Peptisorb)
- II - parenteral glutamine in postoperative time (Active Comparator): The nutritional therapy of group II patients will start post-surgery. It will be based on early enteral nutrition with elementary diet (Peptisorb) with simultaneous parenteral nutrition with two-chamber bag with 480 kcal energetic value and 5.7g of N contained in standard amino acids administered via peripheral veins. Additionally, glutamine (100 ml of Dipeptiven) will be added to the two-chamber bag. The parenteral nutrition will be administered for five days.
  Interventions: Dietary Supplement: Early postoperative enteral nutrition, based on standard elementary diet (Peptisorb); Drug: glutamine
- III - perioperative oral immunonutrition (Active Comparator): Preoperatively, group III patients will be given commercially available oral diet enriched with arginine (Cubitan, 1 package 3 times per day). Additionally, they will be administered commercially available two-chamber bag with 480 kcal energetic value and 5.7g of N in standard amino acids via peripheral access. The duration of pre-operative preparatory phase ranged between 5 and 10 days (8 days on average). Enteral nutrition with commercially available arginine-containing diet (Cubison) will start 20 hours post-surgery at an 8 ml/h flow rate; the rate will be increased gradually, with the volume doubled every 24 hours, up to 100 ml/h and continued for six days. Simultaneously, commercially available two-chamber bags for peripheral access with composition identical to that used preoperatively will be administered via peripheral veins for five days.
  Interventions: Dietary Supplement: oral diet enriched with arginine (Cubitan)
- IV - Perioperative parenteral immunonutrition (Active Comparator): Nutritional therapy of group IV will be based on intravenous preparations. Two-chamber bags with 480 kcal energetic value and 5.7 g of N in standard amino acids will be administered preoperatively. A solution of glutamine (Dipeptiven, 100 ml) and ω3-fatty acids (Omegaven, 100 ml) will be added to the bags. The duration of pre-operative preparatory phase ranged between 5 and 10 days (8 days on average). Enteral nutrition with elementary commercially available diet (Peptisorb) will be begun 20 hours post-surgery; it will be started at an 8 ml/h flow rate and increased gradually, with the volume doubled every 24 hours, up to 100 ml/h. The enteral nutrition will be continued for six days. During the initial five days post-surgery, the patients will be additionally supplemented parenterally via peripheral veins; similarly to the preoperative period, the content of two-chamber bag for peripheral access enriched with glutamine and ω3-fatty acids will be administered for five days.
  Interventions: Dietary Supplement: Early postoperative enteral nutrition, based on standard elementary diet (Peptisorb); Drug: Perioperative parenteral immunonutrition (Dipeptiven, Omegaven)

INTERVENTIONS:
Dietary Supplement: Early postoperative enteral nutrition, based on standard elementary diet (Peptisorb) — Early postoperative enteral nutrition with standard elementary diet (Peptisorb), will start 20 hours post-surgery. The initial flow rate will be 8 ml/h, which will increase gradually, with the volume doubled every 24 hours, up to 100 ml/h. The enteral nutrition wil be continued for six days. During the initial five days post-surgery, the patients will be additionally supplemented parenterally via peripheral veins (commercially available two-chamber bag for peripheral access with 480 kcal of energetic value and 5.7g of N contained in standard amino acids).
  Arms: I - Nutritional therapy only during the postoperative period.; II - parenteral glutamine in postoperative time; IV - Perioperative parenteral immunonutrition
Drug: glutamine — The nutritional therapy of group II patients will start post-surgery. It will be based on early enteral nutrition with elementary diet (Peptisorb) with simultaneous parenteral nutrition with two-chamber bag with 480 kcal energetic value and 5.7g of N contained in standard amino acids administered via peripheral veins. Additionally, glutamine (100 ml of Dipeptiven) will be added to the two-chamber bag. The parenteral nutrition will be administered for five days.
  Arms: II - parenteral glutamine in postoperative time
Dietary Supplement: oral diet enriched with arginine (Cubitan) — Preoperatively, group III patients will be given commercially available oral diet enriched with arginine (Cubitan, 1 package 3 times per day). Additionally, they were administered commercially available two-chamber bag with 480 kcal energetic value and 5.7g of N in standard amino acids via peripheral access. The duration of pre-operative preparatory phase ranged between 5 and 10 days (8 days on average). Enteral nutrition with commercially available arginine-containing diet (Cubison) will start 20 hours post-surgery at an 8 ml/h flow rate; the rate will increase gradually, with the volume doubled every 24 hours, up to 100 ml/h and continued for six days. Simultaneously, commercially available two-chamber bags for peripheral access with composition identical to that used preoperatively will be administered via peripheral veins for five days.
  Arms: III - perioperative oral immunonutrition
Drug: Perioperative parenteral immunonutrition (Dipeptiven, Omegaven) — Nutritional therapy of group IV will based on intravenous preparations. Two-chamber bags with 480 kcal energetic value and 5.7 g of N in standard amino acids were administered preoperatively. A solution of glutamine (Dipeptiven, 100 ml) and ω3-fatty acids (Omegaven, 100 ml) will be added to the bags. The duration of pre-operative preparatory phase ranged between 5 and 10 days (8 days on average). Enteral nutrition with elementary commercially available diet (Peptisorb) will be begun 20 hours post-surgery; it will start at an 8 ml/h flow rate and increased gradually, with the volume doubled every 24 hours, up to 100 ml/h. The enteral nutrition was continued for six days. During the initial five days post-surgery, the patients will be additionally supplemented parenterally via peripheral veins; similarly to the preoperative period, the content of two-chamber bag for peripheral access enriched with glutamine and ω3-fatty acids will be administered for five days.
  Arms: IV - Perioperative parenteral immunonutrition

SUMMARY:
Perioperative immunonutrition in gastric cancer patients can reduce perioperative morbidity and may improve quality of their life. Patients with gastric cancer will be divided into four groups depending on the type of artificial nutrition. Group I (enteral feeding) and II (enteral feeding and parenteral nutrition with glutamine) will be administered nutritional therapy during the postoperative period, group III (oral arginine) and IV (parenteral immunonutrition) patients will be treated nutritionally both prior to and after the surgery. The lymphocytes and their subpopulations, interleukin IL-1B,-6,-23, and the phagocytic, and bactericidal activity of blood platelets will be determined before and after nutritional therapy.

DETAILED DESCRIPTION:
Surgical treatment of gastric cancer is associated with a high risk of perioperative complications. Morbidity of cancer patients increases in concert with the clinical stage of the malignancy. It is postulated that a reduction in perioperative morbidity and improved quality of life of patients with advanced gastric cancer can be achieved by proper preparation to surgery, among others. One of such methods is the implementation of immunostimulating nutritional therapy during the perioperative period.The stage of cancer will be graded according to TNM classification. The patients will be randomly assigned to four clinical groups based on the type of nutritional therapy implemented.

ELIGIBILITY:
Inclusion Criteria:

* gastric cancer

Exclusion Criteria:

* for group III constituted gastric cancer associated with severe gastrointestinal obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2007-03; Primary Completion 2021-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Phagocytic activity of blood platelets in gastric cancer patients. | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Platelet count and phagocytic activity of thrombocytes will be examined twice in each patient. Blood samples for laboratory tests will be drawn prior to surgery and nutritional therapy and 12 days after the surgery. Thrombocyte count will be determined using ADVIA 120 haematological analyser. Phagocytic activity of blood platelets will be determined against Staphylococcus aureus ATCC 6538P bacterial strain. It expresses as the fraction of phagocytizing platelets and the phagocytic index. The fraction of phagocytizing platelets corresponds to the percentage of phagocyting thrombocytes per 1000 consecutive cells of this type. The phagocytic index represents the ratio of phagocytized bacteria per 100 phagocytic platelets.

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Kamocki, MD PhD, Principal Investigator — 2nd Department of General and Gastroenterological Surgery Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

REFERENCES:
- [Result] Noisakran S, Gibbons RV, Songprakhon P, Jairungsri A, Ajariyakhajorn Ch, Nisalak A, Jarman RG, Malasit P, Chokephaibulkit K, Perng GC. Detection of dengue virus in platelets isolated from dengue patients. Southeast Asian J Trop Med Public Health. 2009; 40: 253-262. Mustard JF, Packham MA. Platelet phagocytosis. Sem Haematol 1968; 2: 168-184. Clawson CC, White JG.: Platelet interaction with bacteria. I Reaction phases and effects on inhibitors. Am I Pathol 1971; 65: 367-380. Kemona H, Andrzejewska A, Prokopowicz J, Nowak H, Mantur M. Phagocytic activity of human blood platelets examined by electron microscopy. Folia Haematol Int Mag Klin Morphol Blutforsch 1986; 113: 696-702. Bessler H, Agam G, Diadetti M. Increased protein synthesis by human platelets during phagocytosis of latex particles in vivo. Thromb Diath Haemorrh 1976; 35: 350-357. Tang YQ, Yeaman MR, Selsted ME. Antimicrobial peptides from human platelets. Infect Immun 2002; 70: 6524-6533. Yeaman MR. The role of platelets in antimicrobial host defense. Clin Infect Dis 1997; 5: 951-968. Page CP. Platelets as inflammatory cells. Immunopharmacology 1989; 17: 51-59. Sun B, Li J, Kambayashi J. Interaction between GPIbalpha and FcgammaIIa receptor in human platelets. Biochem Biophys Res Commun 1999; 266: 24-27. Kemona H, Andrzejewska A, Prokopowicz J, Nowak H, Mantur M. Phagocytic activity of human blood platelets examined by electron microscopy. Folia Haematol 1986; 113: 696-702. Nash GF, Turner LF, Scully MF, Kakkar AK. Platelets and cancer. Lancet Oncol 2002; 3: 425-430. Yu Y, Zhou XD, Liu YK, Ren N, Chen J. Platelets promote the adhesion of human hepatoma cells with highly metastatic potential to extracellular matrix protein: involvement of platelets P-selectin and GP IIb-IIIa. J Cancer Res Clin Oncol 2002; 128: 283-287. Kamocki Z, Matowicka-Karna J, Piotrowski Z, Kemona H. Bacteriocidal capacity of platelets in gastric cancer patients. Neoplasma 2004; 51: 265-268
- [Derived] Kamocki Z, Matowicka-Karna J, Gryko M, Zareba K, Kedra B, Kemona H. The effect of perioperative immunonutrition on the phagocytic activity of blood platelets in advanced gastric cancer patients. Clin Dev Immunol. 2013;2013:435672. doi: 10.1155/2013/435672. Epub 2013 Dec 1. PMID 24363760